CLINICAL TRIAL: NCT06325475
Title: Comparison of Patients' Postpartum Recovery Using ObsQoR-10 Score in Pregnant Women in Vaginal Delivery With and Without Neuraxial Labor Analgesia: A Single-center Observational Study.
Brief Title: Comparison of Patients' Postpartum Recovery Using ObsQoR-10 Score in Pregnant Women in Vaginal Delivery With and Without Neuraxial Labor Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Aysenur Dostbil, clinical professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/530
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Pregnant women in Group A will receive neuraxial labor analgesia (dural puncture epidural or combined spino epidural analgesia).
  If postpartum analgesic needs arise, patients in Group A will receive 0.0625% bupivacaine via epidural route.
  Interventions: Procedure: labor with neuraxial labor analgesia
- Group B (Active Comparator): Pregnant women in Group A will not receive neuraxial labor analgesia. If postpartum analgesic needs arise, patients in Group B will receive iboprufen and acetaminophen if needed.
  Interventions: Procedure: labour without noroaxial labor analgesia

INTERVENTIONS:
Procedure: labor with neuraxial labor analgesia — Pregnant women in Group A will receive neuraxial labor analgesia (dural puncture epidural or combined spino epidural analgesia).
  If postpartum analgesic needs arise, patients in Group A will receive 0.0625% bupivacaine via epidural route.
  Arms: Group A
Procedure: labour without noroaxial labor analgesia — Pregnant women in Group B will not receive neuraxial labor analgesia (dural puncture epidural or combined spino epidural analgesia).
  If postpartum analgesic needs arise, patients in Group B will receive iboprufen and acetaminophen.
  Arms: Group B

SUMMARY:
The aim of this study was to compare the postpartum recovery of pregnant women who had vaginal delivery with and without neuraxial labor analgesia using the ObsQoR-10 scoring system.

DETAILED DESCRIPTION:
In this study, we planned to conduct a study to compare the postpartum recovery of pregnant women according to patient-reported outcome measures using the ObsQoR-10 score in vaginal deliveries with and without neuraxial labor analgesia (dural puncture epidural or combined spino epidural analgesia).

In this study, after obtaining the approval of the ethics committee of Atatürk University Faculty of Medicine Hospital and written informed consent of the patients, 40 pregnant women who will deliver vaginally with or without neuraxial analgesia will be prospectively enrolled.

Patients will be randomized by a statistician using a computerized random numbers table and divided into 2 equal groups as Group A and Group B. Pregnant women in Group A will receive neuraxial labor analgesia (dural puncture epidural or combined spino epidural analgesia), while Group B will not. If postpartum analgesic needs arise, patients in Group A will receive 0.0625% bupivacaine via epidural route, while pregnant women in Group B will receive iboprufen and acetaminophen if needed.

ObsQoR-10 scores of the postpartum patients will be evaluated and recorded at discharge. In addition, basic demographic information and medical, analgesic and obstetric parameters related to the peripartum period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥18 years old
* Pregnant women consenting to neuraxial analgesia for labor
* Being ≥37 weeks gestation

Exclusion Criteria:

* Patients in whom neuraxial analgesia is contraindicated
* Being <18 years old
* Being <37 weeks gestation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-26 (Estimated); Primary Completion 2024-07-26 (Estimated); Study Completion 2024-08-26 (Estimated)

PRIMARY OUTCOMES:
ObsQoR-10 scores of postpartum patients | Patients' ObsQoR-10 scores will be determined at 24 hours postpartum
  ObsQoR-10 scores of postpartum patients will be recorded before discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Dostbil, Study Director — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Background] Sultan P, Kormendy F, Nishimura S, Carvalho B, Guo N, Papageorgiou C. Comparison of spontaneous versus operative vaginal delivery using Obstetric Quality of Recovery-10 (ObsQoR-10): An observational cohort study. J Clin Anesth. 2020 Aug;63:109781. doi: 10.1016/j.jclinane.2020.109781. Epub 2020 Mar 20. PMID 32203873
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408